CLINICAL TRIAL: NCT00308672
Title: The Study for the Prevalence of Metabolic Syndrome and Its Associated Factors in an Urban City- Comparison of Agreement for Prevalence of Metabolic Syndrome Among the WHO, NCEP ATP III and Taiwan Definitions
Brief Title: The Prevalence of Metabolic Syndrome and Its Associated Factors in an Urban City
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: NSC94-2314-B-039-024
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2006-03

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The secondary objective is to evaluate the agreement between these criteria and the prevalence of concordant and discordant according to different criteria.

DETAILED DESCRIPTION:
Up to now, there has been to uniform case definition for the metabolic syndrome. The World Health Organization and the Third Report of the National Cholesterol Education Program's Adult Treatment Panel (ATP III), and Bureau of Health Promotion, Taiwan proposed different criteria for the metabolic syndrome. Therefore, the secondary objective is to evaluate the agreement between these criteria and the prevalence of concordant and discordant according to different criteria. Three thousand persons will be randomly selected from resident of Taichung City. All the participants will fulfill a structured questionnaire. Blood pressure, anthropometric variables are measured. Biochemical markers are analyzed by a biochemical autoanalyzer. Kappa will be used to estimate the agreement between different criteria.

ELIGIBILITY:
Inclusion Criteria:

Residents aged 40 and over of Taichung City, Taiwan in October, 2004.

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Lin C Chieh, Professor, Principal Investigator — School of Medicine, China Medical Universtiy
Locations (1):
- China Medical University Hospital, Taichung, Taiwan